CLINICAL TRIAL: NCT03428269
Title: Comparative Value of a Serious Game and a Traditional Teaching Method to Improve Clinical Reasoning Skills Necessary to Detect Patient Deterioration: A Randomized Study in Nursing Students
Brief Title: Serious Game Versus Traditional Teaching to Improve Clinical Reasoning Skills
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université Paris-Sud (Other)
Responsible Party: Principal Investigator, Antonia Blanie, principal investigator, Université Paris-Sud
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: LabForSims-003
Record Dates: First submitted 2018-01-30; First posted 2018-02-09 (Actual); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: Simulation
Keywords: simulation; clinical reasoning; patient deterioration

STUDY DESIGN:
Intervention Model Description: Parallel assignment, not blinded, randomized study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- simulation by gaming group (Experimental): In the simulation by gaming group, the students will individually play with two cases of the LabforGames Warning game (postoperative hemorrhage case and brain trauma in elderly case). After each case, a debriefing to which with all players will participate will be conducted by an instructor.
  Interventions: Other: simulation by gaming (LabForGames Warning)
- traditional education group (Active Comparator): In traditional education group, the students will individually work on the two same cases but the two vignettes and adjoining questions will be presented and answered by the student on a paper sheet. Then a global review of the two cases and the major messages to be retained will be presented by a teacher.
  Interventions: Other: traditional education

INTERVENTIONS:
Other: simulation by gaming (LabForGames Warning) — comparison of the efficacy of two educational methods to improve the clinical reasoning skills of nursing students facing patient deterioration
  Arms: simulation by gaming group
Other: traditional education — comparison of the efficacy of two educational methods to improve the clinical reasoning skills of nursing students facing patient deterioration
  Arms: traditional education group

SUMMARY:
Detection of patient deterioration is a major healthcare problem. Indeed, acute clinical deterioration of the patient is often preceded by changes of several physiological parameters within 6 to 24h before the event occurs. The combination of i) early detection ii) rapid response and iii) efficient clinical management influences the patient's prognosis. Education of nurses, who are frontline healthcare providers, is therefore essential. Serious games might represent an interesting immersive educational tool to train a large number of healthcare professionals with high flexibility but assessment of their learning efficacy should be demonstrated. A serious game named LabforGames Warning has been developed for nursing students with the aims of improving their ability to detect clinical deterioration and to promote adequate interprofessional communication. The objective of this study will be to compare the respective value of digital simulation (using the above mentioned serious game) and a traditional teaching method to improve the clinical reasoning skills necessary to detect patient deterioration.

DETAILED DESCRIPTION:
Detection of patient deterioration is a major healthcare problem. Indeed, acute clinical deterioration of the patient is often preceded by changes of several physiological parameters within 6 to 24h before the event occurs. The combination of i) early detection ii) rapid response and iii) efficient clinical management influences the patient's prognosis. Education of nurses, who are frontline healthcare providers, is therefore essential.

Serious games might represent an interesting immersive educational tool to train a large number of healthcare professionals with high flexibility but assessment of their learning efficacy should be demonstrated. The investigators are interested to explore the relative benefits of gaming over other methods of training and how can non-technical skills be improved by gaming. A serious game named LabforGames Warning has been developed by the investigators with the aims of improving nursing students' capacity to detect patient deterioration and to promote adequate interprofessional communication. It includes four different scenarios in various clinical conditions (postoperative hemorrhage, pediatric diarrhea and hypovolemia, brain trauma in an elderly patient, abdominal occlusion in a psychiatric patient) but in all of them deterioration of the patient status occurs in three consecutive steps (minimal, moderate and severe). Each scenario can be used separately but all can also be played sequentially. The game can be used in a dedicated room with several computers allowing several students to play at the same time (multiplayer format). It can also be played alone by accessing the university website with each student being given a login and a password (single player format). The game conception emphasizes the fact the each student can play the game several times until his (her) score reaches an excellent result. When the game is played in a room of the medical/nursing school with 15-20 students performing at the same time, a common interactive debriefing is provided by an instructor at the end of each scenario in addition to the feedback included in the game itself. A pre-formatted feedback is indeed provided on the screen of the computer at the end of each step of the scenario and emphasizes the major lessons to be understood and retained for this part of the game. When the player uses the serious game alone during an internet-based session, the debriefing is limited to the pre-formatted feedback.

The nursing student is seated in front of the screen of the computer and uses a mouse to move objects and respond to questions. Initially, the player is informed on the clinical environment of the game and technical information (how to manipulate the items on the screen) is provided. Responses provided by the student in the consecutive stages of the scenario are scored (a scoring system has been previously established by the instructors who developed the game) and a feedback explaining the main issues (errors or imperfect responses) is also provided on the computer screen. At each clinical step during a given scenario, the player has the possibility to call a physician but the content of the information provided and the details of the request are examined and scored.

In the present study, the objective will be to compare the respective educational value of the above mentioned serious game and a traditional teaching method to improve the clinical reasoning skills necessary to detect patient deterioration.

This randomized study will be performed in the simulation center of Paris Sud University (LabForSIMS). After informed consent, 2nd year nursing students from nursing schools will be included and randomized into two groups: simulation by gaming group and traditional teaching group (control group).

In the simulation by gaming group, students will individually play with two scenarios of LabforGames Warning (postoperative hemorrhage after hip replacement and brain trauma in an elderly patient).

In the traditional teaching group, an instructor will present and discuss the same two vignettes with a similar number of students (i.e. 15 students). Information is presented using paper and a PowerPoint slide kit. The duration of the course will be similar to that of the serious game session.

The student's clinical reasoning skills will be measured by script concordance tests (SCT) to assess the retention of the clinical reasoning skills. A series of 80 SCT related to the learning objectives of the session will be presented to each group immediately after the session and one month thereafter. In addition, the perceived satisfaction and the effectiveness of the instructional design will be assessed using a questionnaire at the end of the session.

ELIGIBILITY:
Inclusion Criteria:

* nursing students

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
clinical reasoning skills | 20 minutes at the end of the session
  assessed by the global score of script concordance tests (score between 0 to 100)

SECONDARY OUTCOMES:
self efficacy | 1 minutes at end of the session
  measured by a Likert scale between 1 to 10
satisfaction | 1 minutes at end of the session
  measured by a Likert scale between 1 to 10)
retention of clinical reasoning skills | 20 minutes one month after
  assessed by the global score of script concordance tests

CONTACTS AND LOCATIONS:
Overall Officials: Antonia BLANIE, MD, Principal Investigator — Université Paris-Sud
Locations (4):
- France (4):
  - IFSI Sud Francilien, Corbeil-Essonnes
  - IFSI etampes, Étampes
  - IFSI Perray Vaucluse, Sainte-Geneviève-des-Bois
  - IFSI Paul Guiraud, Villejuif

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dory V, Gagnon R, Vanpee D, Charlin B. How to construct and implement script concordance tests: insights from a systematic review. Med Educ. 2012 Jun;46(6):552-63. doi: 10.1111/j.1365-2923.2011.04211.x. PMID 22626047
- [Derived] Blanie A, Amorim MA, Benhamou D. Comparative value of a simulation by gaming and a traditional teaching method to improve clinical reasoning skills necessary to detect patient deterioration: a randomized study in nursing students. BMC Med Educ. 2020 Feb 19;20(1):53. doi: 10.1186/s12909-020-1939-6. PMID 32075641